CLINICAL TRIAL: NCT07070648
Title: Study on Predicting Response to Standard First-Line Treatment in Diffuse Large B-Cell Lymphoma (DLBCL) Patients Using ctDNA Combined With PET: A Prospective, Multicenter, Multicohort Investigation
Brief Title: Study on Predicting Response to Standard First-Line Treatment in Diffuse Large B-Cell Lymphoma (DLBCL) Patients Using ctDNA Combined With PET
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Rong Tao, Professor, Fudan University
Other Study IDs: SHCA-HEMA-03
Record Dates: First submitted 2025-06-24; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Large B-Cell Lymphoma; DLBCL
Keywords: Diffuse Large B-Cell Lymphoma; ctDNA; PET-CT
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma ctDNA detection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pola-R-CHP treatment group (IPI score 2-5): Pola-R-CHP treatment group (IPI score 2-5)
  Interventions: Drug: POLA-R-CHP

INTERVENTIONS:
Drug: POLA-R-CHP — Pola-R-CHP treatment for 6 cycles (IPI score 2-5)

SUMMARY:
This is a prospective, multicenter, multi-cohort study of ctDNA combined with PET for predicting the efficacy of standard first-line therapy for patients with newly diagnosed diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
This multicenter, prospective, multi-cohort clinical study was designed to evaluate the relevance of combined test results for PET / CT and ctDNA and patient survival outcomes in patients with naive DLBCL after 2 cycles of treatment with the standard first-line therapy. The study plans to enroll 80 patients with newly diagnosed, CD20-positive DLBCL who have not received prior systemic therapy. Participants will be stratified into two cohorts based on baseline International Prognostic Index (IPI) scores, receiving either the NMPA-approved R-CHOP regimen (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone) or the NMPA-approved Pola-R-CHP regimen (polatuzumab vedotin, rituximab, cyclophosphamide, doxorubicin, prednisone) for 6 cycles. PET/CT imaging will be performed at baseline, Cycle 2 Day 20 (C2D20), and 6 weeks after Cycle 6 Day 21 (C6D21), while whole-blood samples for circulating tumor DNA (ctDNA) analysis will be collected at baseline, Cycle 3 Day 1 (C3D1), and C6D21.The primary endpoint of this study is the association of PET / CT and ctDNA test results with progression-free survival (PFS) after 2 cycles of RCHOP or Pola-R-CHP regimen in treatment-naive patients with diffuse large B cell lymphoma (DLBCL). Secondary endpoints are the correlation between the combination of PET / CT and ctDNA with tumor remission after 2 cycles of RCHOP or Pola-R-CHP in DLBCL patients, association of PET / CT and ctDNA with RCHOP or Pola-R-CHP and assessment of the CR rate, ORR, EFS and safety of real-world RCHOP or Pola-R-CHP regimen in treatment-naive DLBCL patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Previously untreated CD20-positive DLBCL patients, including the following types according to the 2016 WHO classification of lymphoid neoplasms: DLBCL, not otherwise specified (NOS) including germinal center B-cell type and activated B-cell type; T-cell/histiocyte-rich large B-cell lymphoma; Epstein - Barr virus-positive DLBCL, NOS; ALK-positive large B-cell lymphoma; HHV8-positive DLBCL, NOS; high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements (double-hit or triple-hit lymphoma); high-grade B-cell lymphoma, NOS.
* Signed informed consent form (ICF).
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 - 2, with an expected survival greater than 12 months.
* Have at least one measurable two-dimensional lesion determined by clinical examination, CT scan, or MRI: ① lymph nodes > 1.5 cm; ② other non-lymph node lesions ≥ 1.0 cm.
* Good function of major organs: Hematological function: absolute neutrophil count ≥ 1,000/mm³, platelet count ≥ 75,000/mm³; Liver function: ALT/AST < 3 times the upper limit of normal (ULN) and total bilirubin ≤ 1.5× ULN (for patients with Gilbert syndrome, hilar compressive adenopathy-induced cholestasis, liver involvement or lymphoma-induced biliary obstruction < 5 times ULN); Renal function: creatinine clearance > 30 mL/min, creatinine ≤ 1.5× ULN; Pulmonary function: indoor oxygen saturation ≥ 95%; Cardiac function: no obvious cardiac insufficiency or cardiovascular disease.
* Fertile patients must be willing to take highly effective contraceptive measures during the study and within 120 days after the last administration of treatment.

Exclusion Criteria:

* Patients planned to receive short-cycle chemotherapy and radiotherapy.
* Subjects judged by the investigator to have any factors affecting compliance with the protocol, including uncontrollable medical, psychological, family, sociological or geographical conditions; or unwilling or unable to comply with the procedures required in the study protocol.
* Known human immunodeficiency virus (HIV) infection or positive immunassay.
* Viral infections that cannot be controlled by antiviral drugs, such as herpesvirus active infection, acute or chronic active hepatitis B, acute or chronic active hepatitis C, etc. (Note: Chronic HBV carriers or inactive HBsAg-positive subjects with HBV-DNA below the detection limit can be enrolled, requiring clinical evaluation, and if appropriate, preventive antiviral treatment is required; HCV antibody-negative subjects can be enrolled, and HCV antibody-positive patients need to be tested for HCV-RNA, and if negative, they can be enrolled).
* Patients with uncontrolled lymphoma central nervous system infiltration (central nervous system diseases diagnosed at the initial diagnosis are allowed, provided that complete remission of central nervous system diseases is achieved and maintained and there is no central nervous system disease at recurrence).
* Pregnant or lactating patients.
* Other concurrent serious diseases or medical conditions that would interfere with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed diffuse large B - cell lymphoma (DLBCL)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between combined PET/CT and ctDNA assessments after 2 cycles of R-CHOP or Pola-R-CHP therapy and progression-free survival (PFS) | Baseline, Day 20 of Cycle 2, and 6 weeks after Cycle 6 completion（each cycle is 21 days）
  Deauville criteria (PET), Lugano 2014 (response), ctDNA (Percentage reduction in ctDNA concentration by NGS kit) Progression-free survival (PFS): Defined as the period from the first administration of medication until disease progression or death from any cause.

SECONDARY OUTCOMES:
Correlation between combined PET/CT and ctDNA assessments after 2 cycles of R-CHOP or Pola-R-CHP therapy and tumor response and overall survival (OS) in treatment-naive DLBCL patients | Through study completion, an average of 2 year"
  Real-world evaluation of complete response rate (CRR), overall response rate (ORR), progression-free survival (PFS), event-free survival (EFS), overall survival (OS), and safety profiles of R-CHOP or Pola-R-CHP regimens in treatment-naive diffuse large B-cell lymphoma (DLBCL) patients,ctDNA(positve or negative by NGS kit).

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, M.D, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No